CLINICAL TRIAL: NCT00302055
Title: Feasibility of a Partnered Approach to Prevent Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Ronald Ackermann, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DK71527 (completed)
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-10

CONDITIONS: Pre-diabetic State; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- one-on-one lifestyle (Active Comparator): Clinical referral to diabetes prevention lifestyle intervention at School of Medicine campus
  Interventions: Behavioral: Clinical referral to diabetes prevention lifestyle
- group-based community lifestyle (Experimental): Clinical referral to group diabetes prevention lifestyle intervention program in community
  Interventions: Behavioral: Clinical referral to group diabetes prevention lifestyle

INTERVENTIONS:
Behavioral: Clinical referral to diabetes prevention lifestyle — 16 one-hour lifestyle program sessions (diet and physical activity skill building and problem solving) delivered about once weekly over 20-24 weeks, followed by monthly lifestyle maintenance sessions
  Arms: one-on-one lifestyle
Behavioral: Clinical referral to group diabetes prevention lifestyle — 16 one-hour lifestyle program sessions (diet and physical activity skill building and problem solving) delivered about once weekly over 20-24 weeks, followed by monthly lifestyle maintenance sessions
  Arms: group-based community lifestyle

SUMMARY:
The Diabetes Prevention Program (DPP) demonstrated that an intensive lifestyle intervention resulting in modest weight loss and increased physical activity can delay or prevent the development of type 2 diabetes in those at increase risk for the disease. The lifestyle program used, however, was not designed for delivery on a public health scale. Successful DPP translation will require a sustainable partnership between a health care system and an established community organization committed to community health and experienced in implementing sustainable health and wellness programs. We have been collaborating with local health system and community administrators for over a year to design a 'real-world' clinic-based screening model to identify and refer high-risk patients for a group-based adaptation of the DPP lifestyle intervention in community facilities. We have designed this study to develop preliminary data about the feasibility and yield of clinic-based screening and referral, as well as the effectiveness of the adapted lifestyle intervention. This pilot study seeks to: 1) evaluate the feasibility of a strategy to implement American Diabetes Association (ADA) recommendations for clinic-based diabetes-risk testing and to refer high-risk patients for a community-based lifestyle intervention; 2) compare two strategies to enhance community-based program participation by referred patients; 3) demonstrate the capability of community facilities to schedule and enroll referred clinic patients at high-risk for diabetes and to deliver a modified, group-based DPP lifestyle intervention consistently; and 4) compare levels of weight loss and physical activity achieved by referred clinic patients with pre-diabetes who participate in a free-of-charge, group-based DPP lifestyle intervention at community facilities compared to a free-of-charge, traditional, one-on-one DPP lifestyle intervention at a DPP research site. Addressing these issues now will enable us to evaluate this partnered DPP translation model with a larger, more robust future study that will involve referral by multiple primary care clinics, program delivery at more community sites, and a 3-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

25 years of age or older Body-mass index of >= 24 kg/m2

1. or more additional risk factors if age is <45

   - Parent or sibling with diabetes
   * Minority race or ethnicity
   * History of gestational diabetes
   * Delivery of infant >= 9 lbs.
   * History of high blood pressure
   * History of dyslipidemia
   * Polycystic Ovarian Syndrome
   * History of vascular disease Fasting Capillary Glucose 95 - 125 mg/dl 2-hour Post-challenge Capillary Glucose 140 - 199 mg/dl

   Exclusion Criteria:

   Diseases that could limit lifespan or increase risk with a lifestyle intervention - Cancer diagnosed in the past 5 years

   - Significant Cardiovascular Disease

   - A "Yes" response to any item on the modified Physical Activity Readiness Questionnaire

   - Uncontrolled hypertension: systolic blood pressure >180 mmHg or diastolic blood pressure >105 mmHg
   * Heart attack, stroke, or transient ischemic attack within 6 months
   * Chest pain or unexplained dizziness or fainting with physical exertion
   * Chronic obstructive pulmonary disease or asthma needing home oxygen
   * Other chronic disease or condition, such as advanced arthritis, that could limit ability to become physically active or limit life span to <5 years
   * Any other known reason for not participating in regular physical activity

   Exclusions related to metabolism - Past anti-diabetes medication use, except during gestational diabetes

   - Use of a medications known to produce hyperglycemia

   - Known disease leading to abnormal glucose metabolism

   Exclusions for conditions / behaviors likely to affect study conduct

   - Unable or unwilling to provide informed consent
   * Unable to communicate with the pertinent clinic staff
   * Unable to read written English or Spanish

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald T Ackermann, MD, MPH, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (2):
- United States (2):
  - IU Medical Group Westside Clinic, Indianapolis, Indiana
  - IU Medical Group Banta Road Clinic, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- One-on-one Lifestyle: Clinical referral for diabetes prevention lifestyle intervention at School of Medicine campus
Period: Overall Study
Arm/Group | One-on-one Lifestyle | Group-based Community Lifestyle
Started | 23 | 49
Completed | 14 | 36
Not Completed | 9 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | One-on-one Lifestyle | Group-based Community Lifestyle | Total
Number analyzed (Participants) | 23 | 49 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 49 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (10.7) | 52.8 (13.1) | 52.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 42 | 59
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 23 | 49 | 72

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: We analyzed repeated outcome measures using longitudinal linear regression with 3 observations per participant (baseline, 6 months, and 12 months)
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | One-on-one Lifestyle | Group-based Community Lifestyle
Number analyzed (Participants) | 23 | 49
kilograms | 4.37 [3.33 to 5.42] | 3.23 [2.16 to 4.30]

2. Secondary Outcome: Self Report Physical Activity
Time Frame: 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Rate of Community Program Participation
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse events are solicited from participants at every follow-up measurement time point.
Arm/Group | One-on-one Lifestyle | Group-based Community Lifestyle
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/49
Other Adverse Events (participants affected / at risk) | 0/23 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No